CLINICAL TRIAL: NCT06961123
Title: Establishment of a Longitudinal Cohort for Newborns With Low Apgar Scores at Birth
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BYSYDL2024012
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-03

CONDITIONS: Low Apgar Scores
Keywords: Low Apgar scores, neonatal, birth cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Umbilical cord blood, Meconium
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- At any time after 1 minute, 5 minutes, or 10 minutes of birth, the Apgar score of the newborn is ≤ 7

SUMMARY:
The objective of this study is to identify high-risk factors associated with low Apgar scores, implement proactive interventions to reduce their occurrence, and analyze neonatal resuscitation procedures and systemic treatment during hospitalization. This aims to provide evidence-based references for improving the resuscitation and medical management of newborns with low Apgar scores, thereby enhancing clinical care capabilities. Additionally, continuous follow-up management and timely intervention guidance will be provided to these infants to optimize their long-term prognosis.

DETAILED DESCRIPTION:
This is a prospective and retrospective biphasic cohort study.Retrospective cohort inclusion criteria: Newborns born between January 1, 2006 and before the start of the project at Peking University Third Hospital with Apgar scores ≤ 7 at 1 minute, 5 minutes, or 10 minutes.

Prospective cohort inclusion criteria: Newborns born in our hospital between the start of the project and December 31, 2027, with an Apgar score of ≤ 7 at 1 minute, 5 minutes, or 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Retrospective cohort inclusion criteria: Newborns born between January 1, 2006 and before the start of the project at Peking University Third Hospital with Apgar scores ≤ 7 at 1 minute, 5 minutes, or 10 minutes.

Prospective cohort inclusion criteria: Newborns born at Peking University Third Hospital between the start of the project and December 31, 2027, with an Apgar score of ≤ 7 at 1 minute, 5 minutes, or 10 minutes.

Exclusion Criteria:

* There are serious congenital malformations that affect physical and neurological development, and family members refuse to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborns born at Peking University Third Hospital with Apgar scores ≤ 7 at any time point within 1 minute, 5 minutes, or 10 minutes after birth
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical development indicators, Neurodevelopmental outcome | 6 months old, 1 year old, 2 years old
  Physical development indicators：height, weight, head circumference, BMI, Z-score Neurodevelopmental outcome: Good neural development, poor neural development, cerebral palsy, autism spectrum disorder, Attention deficit hyperactivity disorder

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided